CLINICAL TRIAL: NCT03016156
Title: Determination of the Sensitivity and Specificity of a Smartphone Application to Detect Retinoblastoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Accrual was slow.
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: RBAPP; NCI-2021-05557 (Registry Identifier: NCI)
Record Dates: First submitted 2016-12-28; First posted 2017-01-10 (Estimated); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Retinoblastoma; Cataracts Infantile; Glaucoma, Congenital; Leucocoria
MeSH Terms: conditions — Retinoblastoma; Hydrophthalmos

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stratum I: Initial Evaluation Group (Experimental): Initially, a small group of patients diagnosed with congenital or infantile cataracts, congenital glaucoma or retinoblastoma and who meet the eligibility criteria will undergo testing with CRADLE on Day 1.
  Interventions: Other: CRADLE
- Stratum II: Leukocoria Evaluation Group (Experimental): A separate group of participants who are referred for evaluation of leukocoria or any other eye condition will undergo red reflex testing testing with CRADLE on Day 1.
  Interventions: Other: CRADLE; Other: Red reflex testing
- Stratum III: Retinoblastoma Group (Experimental): A separate group of participants with known retinoblastoma and who are undergoing ocular salvage treatments will be screened with red reflex testing using direct ophthalmoscopy on Day 1. They will also undergo testing with the CRADLE software application defined as the most effect in Stratum I on Day 1 then for three additional consecutive visits which typically occur every 3 to 4 weeks.
  Interventions: Other: CRADLE; Other: Red reflex testing

INTERVENTIONS:
Other: CRADLE — A smartphone software application designed to detect leukocoria using a sophisticated photoluminic analysis.
  The investigator or designee will perform tests with CRADLE in separate patient cohorts with known diagnosis of retinoblastoma, congenital glaucoma, or cataracts.
  Other Names: Smartphone application; ComputeR Assisted Detection of LEukocoria
Other: Red reflex testing — Traditional red reflex testing for leukocoria using a direct ophthalmoscope on routine eye examination. Red reflex testing via direct ophthalmoscope will be performed before dilation, using the ophthalmoscope held close to the examiner's eye, focused on the pupil, viewed at 12 to 18 inches from the patient's eyes, with the room lights dimmed, in accordance with the American Academy of Pediatrics guidelines.
  Other Names: Ophthalmoscopic exam
  Arms: Stratum II: Leukocoria Evaluation Group; Stratum III: Retinoblastoma Group

SUMMARY:
This study seeks to determine whether a smartphone application called CRADLE (ComputeR Assisted Detection of LEukocoria) has the potential to improve the detection of leukocoria. There will be no impact on participants' health outcome.

This study will be performed in two parts, each with a distinct cohort of patients.

Part 1 will assess the feasibility of various techniques/conditions for using CRADLE within patients known to have leukocoria.

Part 2 will estimate the sensitivity and specificity of CRADLE to detect leukocoria (using the techniques selected from information gathered in Part 1) as compared to an ophthalmoscope, within patients referred to the clinic for suspected leukocoria.

PRIMARY OBJECTIVES:

* To determine the most effective usage of a camera phone application (CRADLE) to maximize detection of leukocoria in patients with retinoblastoma, congenital cataracts, and glaucoma.
* To estimate the sensitivity and specificity of a camera phone application (CRADLE) in detecting leukocoria.

DETAILED DESCRIPTION:
This study will utilize three strata called Stratum I, Stratum II and Stratum III.

STRATUM I - Infants and children known to have leukocoria who have been diagnosed with retinoblastoma, cataracts or glaucoma or other eye conditions.

Participants enrolled on Stratum I of the study will have the CRADLE application used by the doctor during their appointment.

The participant will look straight forward while the doctor stands about 1-3 feet away holding the device that has the CRADLE application. He or she will slowly move the device up, down, middle, right, and left - both in a lit and dimmed room.

The participant will be videotaped and photographed during this appointment. The doctor will record the results as determined by CRADLE ("normal" or no leukocoria versus "abnormal" or positive for leukocoria).

STRATUM II - Infants and children who are referred to an eye doctor to evaluate for leukocoria.

Participants enrolled on Stratum II of the study will be asked to look straight forward while he or she uses the CRADLE application (using the best method determined from Stratum I). The doctor will also examine the participant's eyes with the ophthalmoscope method. The results from both CRADLE and the ophthalmoscope method will be recorded and compared (white eye present versus absent, and normal versus abnormal as described above).

STRATUM III - Infants and children receiving treatment for retinoblastoma. For participants enrolled on Stratum III, he or she will have the same procedures as described in Stratum II.

After receiving informed consent, participants will undergo evaluation by ophthalmoscope and CRADLE on Day 1. Stratum III participants only will also undergo CRADLE evaluation on Days 2, 3, and 4.

ELIGIBILITY:
Inclusion Criteria - Stratum I:

* Patient has been diagnosed with congenital or infantile cataracts, congenital glaucoma, or retinoblastoma, and is scheduled for a visit with an ophthalmologist at St. Jude Children's Research Hospital or University of Tennessee Hamilton Eye Institute.
* Patient with retinoblastoma is newly diagnosed, or has received < 2 cycles of chemoreductive therapy, and has not undergone enucleation.
* Patient with cataracts or glaucoma has not received any prior therapy.

Inclusion Criteria - Stratum II:

* Patient without prior diagnosis has been referred for ophthalmological evaluation, including leukocoria or other conditions.

Inclusion Criteria - Stratum III:

* Patient with retinoblastoma undergoing ocular salvage treatment.

Exclusion Criteria

* Prior treatment for cataracts or glaucoma
* Inability or unwillingness of research participant or legal guardian to consent.

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Rate of detection of leukocoria using CRADLE | Day 1
  This outcome will assess the feasibility of various techniques and conditions for using CRADLE in participants with retinoblastoma, congenital cataracts, and glaucoma. The most effective usage of CRADLE to maximize detection of leukocoria will be determined by review of all images, and the most effective and efficient technique will be selected based on the findings and the clarity of the images. This technique will be used for completion of the subsequent objectives using a new cohort of participants.
Sensitivity of CRADLE versus ophthalmoscope to detect leukocoria | Up to Day 4
  The test results obtained by CRADLE will be compared to those obtained by ophthalmoscopic examination to determine the effectiveness of detection of leukocoria by CRADLE. The results will be reported as number of true positive. An ideal test for sensitivity has no false positives.
Specificity of CRADLE versus ophthalmoscope to detect leukocoria | Up to Day 4
  The test results obtained by CRADLE will be compared to those obtained by ophthalmoscopic examination to determine the effectiveness of detection of leukocoria by CRADLE. The results will be reported as number of false negatives (specificity). An ideal test for sensitivity has no false negatives.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Rodriguez-Galindo, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols